CLINICAL TRIAL: NCT06630624
Title: INJECTABL-II: Dose Finding, Efficacy and Immunological Response of a Novel Immuno-Adjuvant (IP-001) Following Microwave Ablation or Irreversible Electroporation for Colorectal Liver Metastases.
Brief Title: Dose Finding, Efficacy and Immunological Response of IP-001 Following MWA or IRE for CRLM
Acronym: INJECTABL-II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.R. Meijerink (Other)
Collaborators: Immunophotonics, Inc. (Industry); Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, M.R. Meijerink, Prof. dr., Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024.0610; 2023-504572-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-06; First posted 2024-10-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Liver Metastases; Liver Metastasis Colon Cancer
Keywords: Colorectal liver metastases; Colorectal hepatic metastases; irreversible electroporation; Microwave ablation; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-dihydrogalactochitosan

STUDY DESIGN:
Intervention Model Description: Firstly, a phase 1, dose-escalation study according to a classic '3+3' design will be performed to determine the maximum tolerated dose (MTD) of intra-tumoral IP-001 injection following MWA. In phase 2 part 1, a single arm study will be performed with the optimal dose found in phase 1 to assess efficacy of intra-tumoral IP-001 injection following MWA in patients with CRLM who will receive the ablation for curative intent. Phase 2 part 2 will be conducted in parallel to phase 2 part 1 as a randomized, two-armed study assessing the efficacy and immunomodulation of intra-tumoral IP-001-injection following two ablative modalities (arm A (MWA) or arm C (IRE)) in patients with refractory metastatic CRC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1 Dose esclatation of IP-001 (Experimental): Intra-tumoral injection of IP-001 following MWA of two pre-defined colorectal liver metastases (CRLM). Patients will receive sequentially higher doses of the IP-001, always divided equally over the two CRLM, regardless of size. Starting dose will be 8 mL and the dose-escalating steps will be 4 mL up to a total of 16 mL per patient.
  Interventions: Drug: IP-001
- Phase 2 Part 1 MWA + IP-001 (Experimental): One to three colorectal liver metastases (CRLM) will be treated with MWA followed by intra-tumoral injection of IP-001.
  Interventions: Drug: IP-001
- Phase 2 part 2 MWA + IP-001 (Experimental): One to four colorectal liver metastases (CRLM) will be treated with MWA followed by intra-tumoral injection of IP-001.
  Interventions: Drug: IP-001
- Phase 2 part 2 IRE + IP-001 (Experimental): One to four colorectal liver metastases (CRLM) will be treated with IRE followed by intra-tumoral injection of IP-001.
  Interventions: Drug: IP-001

INTERVENTIONS:
Drug: IP-001 — Intra-tumoral injection of IP-001 following ablation (MWA or IRE).

SUMMARY:
The primary objectives of this phase I/II, prospective clinical trial, are to assess the optimal dose, efficacy, safety and immunological effect of ablation and intra-tumoral injection of a novel immuno-adjuvant (IP-001) for colorectal liver metastases (CRLM). The study consists of three parts, devided into two phases.

Phase 1 is a dose-escalation study according to a classic '3+3' design, to identify the dose level at which IP-001 exhibits an acceptable level of toxicity following microwave ablation (MWA) of CRLM in refractory metastatic colorectal cancer (CRC) patients.

Phase 2, part 1 and part 2 are performed simultaneously. In phase 2 part 1, a single arm study assesses the efficacy of IP-001 following MWA for CRLM for curative intent. In phase 2 part 2, a randomized, two-armed study assesses the efficacy and immunomodulation of IP-001 following two ablative modalities: arm A (MWA) and arm C (irreversible electroporation (IRE)) for CRLM in refractory metastatic CRC patients.

DETAILED DESCRIPTION:
Rationale: As ablative therapies lead to in situ availability of ablated tumor material, MWA and IRE have been shown to trigger an anti-tumor immune response. However, the magnitude of this response seems insufficient to induce a detectable abscopal effect (shrinkage or disappearance of distant, untreated tumors). In recent years, there has been a growing interest in exploring the potential synergy between ablative techniques and immune activating strategies to induce a more robust, long-term, systemic anti-tumor immune response.

A novel immuno-adjuvant (IP-001) has been developed to address this synergy and trigger a tumor-specific systemic immune response when exposed to liberated tumor antigens following tumor ablation. 1.0% IP-001 for Injection (IP-001) is injected in and around the ablation zone immediately following ablation. IP-001 creates a depot of released tumor antigens after ablation and drives a potent downstream adaptive immune response against these antigens.

The combination of IP-001 with an ablative treatment in patients with CRLM could prove beneficial in terms of improved (distant) progression free survival (PFS) and possibly OS.

Study design: The INJECTABL-II trial is a phase I-II, prospective clinical trial. The primary conducting center will be the Amsterdam UMC (Amsterdam, the Netherlands). The purpose of this trial is to assess the optimal dose, efficacy, safety and immunological effect intra-tumoral injection of IP-001 following ablation. The trial consists of three study parts, divided into two phases. In phase 1 a dose-finding study will be conducted followed by two parallel phase 2 studies, called phase 2 part 1 and phase 2 part 2.

The investigators will first conduct a phase 1, dose-escalation study according to a classic '3+3' design to determine the maximum tolerated dose (MTD) of intra-tumoral IP-001 injection following MWA. In phase 2 part 1, a single arm study will be performed with the optimal dose found in phase 1 to assess efficacy of intra-tumoral IP-001 injection following MWA in patients with CRLM who will receive ablation for curative intent. The investigators hypothesize that MWA + IP-001 is superior to MWA alone in terms of 1-year distant progression-free survival (DPFS). 1-year DPFS will be compared to a matched historical, prospective cohort of the COLLISION trial, in which 126 patients have been included. For the sample size calculation, the one-sided Z-Test with pooled variance has been used, yielding 59 patients to be included in this phase of the trial (MWA + IP-001). Phase 2 part 2 will be conducted in parallel as a randomized, two-armed study assessing the efficacy and immunomodulation of intra-tumoral IP-001-injection following three ablative modalities (arm A (MWA) or arm C (IRE)) in patients with metastatic CRC. Efficacy of each randomized study arm will be assessed independently, and thus a single-group design has been used for the sample size calculations. The study treatment is considered effective when a DCR of 25% is reached at 16 weeks. A one-sided, one-sample Z-test has been used to estimate the standard deviation. Bonferroni correction is used to correct for multiple comparisons. 21 patients per study arm (arm A (MWA) and arm B (IRE)) will be randomized in phase 2 part 2 of the trial.

Study population: : In phase 1 of the trial, patients with metastatic CRC and at least 2 CRLM (1-3 cm) that have received at least 1 line of systemic therapy will be included. In phase 2 part 1 of the trial, patients with 1-3 CRLM (≤3 cm), who will receive MWA for curative intent will be included. In phase 2 part 2 of the trial, patients with refractory, liver only or liver dominant, metastatic CRC, limited extra-hepatic disease and 1-4 CRLM (≤3 cm) eligible for MWA and IRE will be included.

Intervention: All patients will receive ablation and intra-tumoral injection of IP-001 of CRLM. During phase 1, 2 CRLM will be treated with intra-tumoral injection of IP-001 following MWA. During phase 2 part 1, 1-3 CRLM eligble for MWA with curative intent will be treated with intra-tumoral injection of IP-001 following MWA. During phase 2 part 2, 1-4 CRLM will be treated with intra-tumoral injection of IP-001 following MWA or IRE.

ELIGIBILITY:
All phases:

Inclusion Criteria:

* Measurable metastatic CRC based on RECIST v1.1;
* The primary tumor has been resected before study inclusion or the patient is asymptomatic with respect to the in situ primary tumor;
* Last imaging ≤ 4 weeks prior to the on-study ablative procedure;
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of no more than 1;
* A life expectancy of at least 3 months at the time of inclusion;
* Adequate bone marrow, liver, and renal function as assessed by laboratory tests. These results should be judged by the local investigator and should be conducted within 7 days prior to definite inclusion;
* Written informed consent.

Exclusion Criteria:

* Compromised liver function defined as warning signs of portal hypertension, INR > 1,5 without use of anticoagulants, bilirubin > x 1.5 Upper limit of normal range (ULN) ASAT >5.0 x ULN, ALAT >5.0 x ULN.
* Compromised kidney function defined as eGFR <45 ml/min (using the Cockcroft Gault formula);
* Active autoimmune disease requiring disease-modifying therapy at the time of screening or during the study period: i.e. > 10 mg prednisolone per day or other immunosuppressive therapy (e.g. methotrexate);
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results;
* Known allergic reaction to shellfish, crabs, crustaceans, or any trial components;
* Known history of HIV or active Hepatitis C or Hepatitis B infection;
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0); requiring antibiotics;
* Pregnant or breast-feeding subjects; Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment;
* Known allergy to contrast agent that cannot be adequately prevented;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study;
* Major surgery or radiotherapy ≤ 3 weeks (7 days for single fraction of palliative radiotherapy) prior to the on-study ablative procedure;
* Systemic therapy ≤ 4 weeks prior to the on-study ablative procedure;
* CTCAE Grade ≥1 from all side effects of prior therapies or prior procedures at the time of inclusion.

Phase 1

Inclusion Criteria:

* Progressive or stable metastatic CRC on CT-scan after at least 1 lines of standard of care systemic treatment. Standard of care systemic treatment will be defined and determined by the treating oncologist. A summary of standard of care systemic treatment for CRLM as used by the medical oncologists at Amsterdam UMC has been listed in Table 1. Patients can also be included if systemic treatment has to be terminated due to toxicity or when patients refuse (further) systemic treatment, or when patients are in a therapy break from systemic therapy as patients can continue with further systemic treatment one month after the study treatment;
* At least 2 CRLM eligible for MWA with a minimum diameter of 1cm and a maximum diameter of 3cm and one (optional but not required) CRLM that will be left untreated and is eligible for biopsy;
* No limitations on intrahepatic or extrahepatic disease;

Exclusion Criteria:

- No additional exclusion criteria.

Phase 2 part 1:

Inclusion Criteria:

* At least one CRLM and a maximum of three CRLM size ≤ 3 cm eligible for MWA with curative intent;
* Additional unablatable CRLM should be resectable with a maximum of 10 additional CRLM;
* Resectability and ablatability should be re-confirmed intra-operatively by US in case of combined/staged resection and ablation. Intra-operatively also full exploration for hepatic, peritoneal and regional lymph node metastases should be performed;

Exclusion Criteria:

* Radical treatment unfeasible or unsafe (e.g. insufficient FLR);
* The presence of extrahepatic nodal or non-nodal metastases. One locally treatable lung metastasis is allowed;
* Any surgical resection or focal ablative liver therapy for CRLM prior to inclusion;

Phase 2 part 2:

Inclusion Criteria:

* Liver only or liver dominant measurable metastatic CRC based on RECIST v1.1;
* Liver dominant metastatic disease is defined as the hepatic tumorload (number and estimated volume) exceeding the extrahepatic tumorload, with a maximum of 5 unequivocal extrahepatic metastases in ≤2 different organ systems;
* At least 2 CRLM, of which at least one is eligible for the study treatment (RFA, MWA and IRE);
* At least 50% (number and estimated volume) of the CRLM should be eligible for ablation. A maximum of 4 CRLM can be assigned for the study treatment. One CRLM has to be left untreated;
* At least one untreated CRLM and one 'to-be-treated' CRLM should be eligible for biopsy;
* Maximum size of CRLM for study treatment is 3cm;
* Any CRLM with a maximum lesion size of 5cm at time of inclusion;
* Limited extrahepatic disease, restricted to the lungs and lymph nodes, with a maximum lesion size of 3cm at time of inclusion. See below for additional information regarding pulmonary nodules;
* Progressive disease on CT-scan after standard of care systemic treatment. Standard of care systemic treatment will be defined and determined by the treating oncologist. Patients can also be included if systemic treatment has to be terminated due to toxicity or when patients refuse (further) systemic treatment.;

Exclusion Criteria:

* Tumor diameter of ≥ 5 cm of any hepatic lesion at the time of inclusion. If lesion size exceeds 5 cm at start of the procedure, the patient will not be excluded;
* Metastases in the lungs or lymph nodes ≥ 3 cm. If lesion size exceeds 3 cm at start of the procedure, the patient will not be excluded;
* Metastases in any other organ than the liver, lungs of lymph nodes;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Phase 1) | During the 10-day DLT-monitoring period.
  The highest dose of IP-001 that does not cause unacceptable side effects defined as the dose level below the dose level that caused 2 or more Dose Limiting Toxicites (DLTs).
1-Year Distant Progression Free Survival (DPFS) (Phase 2 part 1) | 1 year
  Overall DPFS is defined as the time from inclusion to the time of disease progression (according to the RECIST 1.1 guideline) or death (events). Death related to other causes is considered a failure event for DPFS.
Disease Control Rate (DCR) (Phase 2 part 2) | 16 weeks
  DCR is calculated as the percentage of patients experiencing either iSD (Stable Disease), iPR (Partial Response) or iCR (Complete Response) as best response in target lesions at 16 weeks after treatment according to iRECIST.

SECONDARY OUTCOMES:
Elimination half-life of the study drug IP-001 in the blood (t1/2 ) (Phase 1 and phase 2 part 2) | Prior to and +1 hour, +2 hours, +6 hours, +12 hours and + 24 hours after study treatment
  Blood samples will be taken prior to and at different timepoints after the procedure for pharmacokinetic analysis defined as elimination half-life of the study drug IP-001 in the blood.
Overall Survival (OS; per patient analysis) (All phases) | Up to 5 years
  OS is defined as the time from focal therapy to the time of death due to any cause, assessed up to 5 years;
(Serious) Adverse Events ((S)AEs) (All phases) | Up to 5 years
  (Serious) adverse events according to CTCAE v5.0, assessed up to 5 years.
Duration of best overall response (DoR, per patient analysis) (Phase 2 part 2) | Up to 3 years
  DoR is defined from when the time measurement criteria are first met for CR/iCR or PR/iPR until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years;
Local Tumor Progression Free Survival (LTPFS, per lesion analysis) (All phases) | Up to 5 years
  LTPFS is defined as the time from focal therapy to the time of local tumor progression or death from any cause, whichever occurs first. Local tumor is defined as the treated tumor, assessed up to 5 years.
Distant Progression Free Survival (DPFS; per patient analysis) (All phases) | Up to 5 years
  DPFS is defined as the time from focal therapy to the time of distant disease progression or death from any cause, whichever occurs first, assessed up to 5 years. Distant disease is defined as extra-hepatic lesions and untreated, hepatic lesions;
Hepatic progression free survival (HPFS; per patient analysis) (All phases) | Up to 5 years
  HPFS is defined as the time from focal therapy to the time of progression of any tumor in the liver (treated or untreated) or death from any cause, whichever occurs first, assessed up to 5 years;
Time to progression (TTP; per patient analysis) (All phases) | Up to 5 years
  TTP is defined as the time from focal therapy to the time of unequivocal disease progression (events); the date of death from any cause or death without established RECIST progressive disease is considered to be a competing risk. TTP will be analysed with and without competing risks. Assessed up to 5 years.
Progression-free survival (PFS; per patient analysis) (All phases) | Up to 5 years
  The time until the date of unequivocal disease progression (local site recurrence or metastatic disease) or death from any cause, whichever occurs first, assessed up to 5 years.
Disease-free survival (DFS; per patient analysis) (All phases) | Up to 5 years
  DFS is defined as the time from focal therapy until the appearance or worsening of signs or symptoms of the disease or death from any cause, whichever occurs first, assesed up to 5 years.
Pain assessment (Per procedure analysis) | Up to 1 year
  Pain assessment using visual analogue scale questionnaires (VAS; per procedure analysis). Assessed prior to, directly after and every three months after local treatment, and up to 1 year.
Ablative Success (All phases) | Directly after treatment
  Ablative success (or technical success rate) is defined as the primary efficacy rate; the percentage of successfully eradicated tumor tissue after the local treatment, assessed directly after the treatment.
Quality of Life using EORCT QLQ-C30 questionnaireS (QoL; per patient analysis) (Phase 2) | 1 year
  The quality of life is assessed using EORCT QLQ-C30 questionnaires, prior to, and every three months after treatment during a total follow-up time of 1 year.
Quality of Life using EQ-5D questionnaires (QoL; per patient analysis) (Phase 2) | 1 year
  The quality of life is assessed using EQ-5D questionnaires, prior to, and every three months after treatment during a total follow-up time of 1 year.
Quality of Life using PRODISQ questionnaires(QoL; per patient analysis) (Phase 2) | 1 year
  The quality of life is assessed using PRODISQ questionnaires, prior to, and every three months after treatment during a total follow-up time of 1 year.
Time of maximum observed concentration of the study drug IP-001 in the blood (Tmax) (Phase 1 and phase 2 part 2) | Prior to and +1 hour, +2 hours, +6 hours, +12 hours and + 24 hours after study treatment
  Blood samples will be taken prior to and at different timepoints after the procedure for pharmacokinetic analysis defined as time of maximum observed concentration of the study drug IP-001 in the blood.
Maximum observed concentration of the study drug IP-001 in the blood (Cmax) (Phase 1 and phase 2 part 2) | Prior to and +1 hour, +2 hours, +6 hours, +12 hours and + 24 hours after study treatment
  Blood samples will be taken prior to and at different timepoints after the procedure for pharmacokinetic analysis defined as maximum observed concentration of the study drug IP-001 in the blood.
Area under the curve from time 0 to the time of the last measurable concentration of the study drug IP-001 in the blood (AUC 0-t) (Phase 1 and phase 2 part 2) | Prior to and +1 hour, +2 hours, +6 hours, +12 hours and + 24 hours after study treatment
  Blood samples will be taken prior to and at different timepoints after the procedure for pharmacokinetic analysis defined as the area under the curve from time 0 to the time of the last measurable concentration of the study drug IP-001 in the blood.

OTHER OUTCOMES:
Immunomodulation in tissue biopsies (Phase 1 and phase 2 part 2) | Prior to the procedure and 4 weeks post-procedure.
  The effect on treated and untreated tumor tissue will be assessed by pre- and post-treatment biopsies of treated and untreated tumor tissue. The pre- and post-treatment biopsies will be compared to determine the evidence for the induction of a sustainable, infiltrative immune response. Tissue biopsies from the untreated metastasis will be used to investigate the possible induction of a systemic immune response;
Immunomodulation in circulating immunecells (Phase 1 and phase 2 part 2) | prior to the study procedure and +1 day, +10 days, +4 weeks and +8 weeks after the study procedure
  The effect on circulating immune cells and a possible induction of a systemic anti-tumor immune response will be assessed by taking pre- and post-treatment venous blood samples. Samples will be taken prior to the study procedure and after the study procedure after 1 day, 10 days, 4 weeks and 8 weeks.
Effect on circulating tumor DNA (ctDNA) (Phase 2 part 1) | 1 year
  CtDNA is samples to monitor the efficacy of the study treatment (MWA + IP-001), defined as a significant decrease in ctDNA, as well as to predict (radiological) metastatic recurrence or progression, defined as a significant increase in ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn R. Meijerink, Prof., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC - location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No